CLINICAL TRIAL: NCT06019676
Title: Impact of Apalutamide in Metastatic Hormone Sensitive Prostate Cancer Patients, a Multicentre Prospective Observational Study
Brief Title: Impact of Apalutamide in Metastatic Hormone Sensitive Prostate Cancer Patients
Acronym: ADAPT-P
Status: Active, not recruiting | Type: Observational
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Collaborators: Janssen, LP (Industry)
Responsible Party: Sponsor
Other Study IDs: CCR5793
Record Dates: First submitted 2023-08-17; First posted 2023-08-31 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Metastatic Hormone-Sensitive Prostate Cancer (mHSPC)

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients with mHSPC and treatment decision for apalutamide by clinician

SUMMARY:
The ADAPT study is an observational study of apalutamide, which can be given to patients with hormone sensitive metastatic prostate cancer as standard of care. The clinical decision for patients to have apalutamide as part of their management plan will be decided by the clinician. The patient will only be approached about the ADAPT study if they decide they want to have apalutamide as part of their management.

The aims of the ADAPT study include documenting the biochemical effectiveness, as determined by the Prostate-Specific Antigen (PSA) and impact of apaluatmide on health related quality of life. The blood test for PSA is regularly monitored as standard of care.

Additionally, the impact of apalutamide on fatigue, cognitive function, patients reported outcomes, health related quality of life will be evaluated using patient questionnaires answered at defined timepoints. The questionnaires will be sent either electronically or via post at week 12, 24, 36, 48, 72 and 104 weeks after commencement of apalutamide.

Currently, the majority of data regarding tolerability and biochemical response to apalutamide has been from large phase III trials, where there are strict eligibility criteria. Real-world data as from the ADAPT study can provide valuable complementary data to randomised controlled trials, which can be used to address the 'generalizability' limitations of randomised control trials and can provide evidence on the external validity of their findings. This information can advance knowledge of patterns of care, treatment effectiveness and side-effects and inform clinical practice to improve outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Male 18 years of age or older
* Histologically confirmed diagnosis of adenocarcinoma of the prostate with both:
* Metastatic hormone sensitive prostate cancer
* Treatment decision for apalutamide by clinician

Exclusion Criteria:

* Non-metastatic prostate cancer
* Prior chemotherapy / abiraterone / apalutamide / darolutamide / enzalutamide for prostate cancer
* Unable to complete patient reported outcome questionnaires

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Males 18 years of age or older, with metastatic hormone sensitive prostate cancer
Sampling Method: Non-Probability Sample
Enrollment: 170 (Actual)
Dates: Start 2023-09-26 (Actual); Primary Completion 2027-04-01 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
Undetectable PSA rate (defined as PSA <0.2ng/ml by end of year 1 and year 2) in mHSPC patients receiving apalutamide | August 2023 - April 2027

SECONDARY OUTCOMES:
The impact of apalutamide on fatigue, assessed using patient-reported Brief Fatigue Inventory questionnaire | August 2023 - April 2027
The impact of apalutamide on cognitive function, using patient-reported FACT-Cog questionnaire | August 2023 - April 2027
The impact of apalutamide on health-related quality of life, using patient-reported EQ-5D-5L questionnaire | August 2023 - April 2027

OTHER OUTCOMES:
Health care professional experience on the use of apalutamide, assessed using Health Care Professional Questionnaire | August 2023 - April 2027

CONTACTS AND LOCATIONS:
Overall Officials: Julia Murray, Dr., Principal Investigator — The Royal Marsden Hospital, NHS Foundation Trust
Locations (12):
- United Kingdom (12):
  - The Royal Marsden Hospital, Sutton, Surrey
  - Buckinghamshire Healthcare NHS Trust, Aylesbury
  - Northern Ireland Cancer Centre, Belfast Health & Social Care Trust, Belfast
  - East Lancashire Hospitals NHS Trust, Blackburn
  - Addenbrooke's Hospital, Cambridge University Hospitals NHS Foundation Trust, Cambridge
  - Velindre Cancer Centre, Velindre University NHS Trust, Cardiff
  - University Hospitals of Morecambe Bay NHS Foundation Trust, Lancaster
  - Clatterbrdige Cancer Centre, NHS Foundation Trust, Liverpool
  - The James Cook University Hospital, South Tees Hospitals NHS Foundation Trust, Middlesbrough
  - South Tyneside and Sunderland NHS Foundation Trust, Newcastle
  - Freeman Hospital, The Newcastle upon Tyne Hospitals NHS Foundation Trust, Newcastle
  - The University Hospital of North Tees, Stockton-on-Tees

IPD SHARING:
Plan to Share IPD: No